CLINICAL TRIAL: NCT05596110
Title: Acute Effects of Transcutaneous Electrical Nerve Stimulation and Kinesio Taping on Lower Limb Joint Proprioception, Static Standing Balance, Limits of Stability and Functional Balance Performance in Community-dwelling Older Adults
Brief Title: TENS and Taping for Older People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shirley S.M. Fong, Principal Investigator, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CU1
Record Dates: First submitted 2022-10-15; First posted 2022-10-27 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Postural; Defect
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TENS and KT (Experimental): TENS will be applied on the medial and lateral joint lines of the knee and ankle joints and the anterior and posterior joint lines of the hip joint of both legs. In addition, KT will be applied to major postural muscles including the bilateral gluteus medius, quadriceps, and gastrocnemius of the participants.
  Interventions: Behavioral: TENS and KT
- TENS and sham taping (Sham Comparator): TENS will be applied on the medial and lateral joint lines of the knee and ankle joints and the anterior and posterior joint lines of the hip joint of both legs. In addition, sham tapes will be applied to major postural muscles including the bilateral gluteus medius, quadriceps, and gastrocnemius of the participants.
  Interventions: Behavioral: TENS and sham taping
- KT and sham TENS (Sham Comparator): KT will be applied to major postural muscles including the bilateral gluteus medius, quadriceps, and gastrocnemius of the participants. In addition, sham TENS will be applied on the medial and lateral joint lines of the knee and ankle joints and the anterior and posterior joint lines of the hip joint of both legs.
  Interventions: Behavioral: KT and sham TENS
- Sham TENS and sham taping (Sham Comparator): Sham TENS will be applied on the medial and lateral joint lines of the knee and ankle joints and the anterior and posterior joint lines of the hip joint of both legs. In addition, sham tapes will be applied to major postural muscles including the bilateral gluteus medius, quadriceps, and gastrocnemius of the participants.
  Interventions: Behavioral: Sham TENS and sham taping

INTERVENTIONS:
Behavioral: TENS and KT — TENS will be delivered using three E704SD TIMER TENS devices (or similar) through pairs of electrodes placed on the medial and lateral joint lines of the knee and ankle joints and the anterior and posterior joint lines of the hip joint of both legs. In addition, KT (Kinesio Tex Gold) will be applied to major postural muscles including the bilateral gluteus medius (i.e., crosses hip joint), quadriceps (i.e., crosses the knee joint), and gastrocnemius (i.e., crosses ankle joint) of the participants.
  Arms: TENS and KT
Behavioral: TENS and sham taping — TENS will be delivered using three E704SD TIMER TENS devices (or similar) through pairs of electrodes placed on the medial and lateral joint lines of the knee and ankle joints and the anterior and posterior joint lines of the hip joint of both legs. In addition, sham tapes will be applied to major postural muscles including the bilateral gluteus medius (i.e., crosses hip joint), quadriceps (i.e., crosses the knee joint), and gastrocnemius (i.e., crosses ankle joint) of the participants.
  Arms: TENS and sham taping
Behavioral: KT and sham TENS — KT (Kinesio Tex Gold) will be applied to major postural muscles including the bilateral gluteus medius (i.e., crosses hip joint), quadriceps (i.e., crosses the knee joint), and gastrocnemius (i.e., crosses ankle joint) of the participants. In addition, sham TENS will be applied on the medial and lateral joint lines of the knee and ankle joints and the anterior and posterior joint lines of the hip joint of both legs.
  Arms: KT and sham TENS
Behavioral: Sham TENS and sham taping — Sham TENS will be applied on the medial and lateral joint lines of the knee and ankle joints and the anterior and posterior joint lines of the hip joint of both legs. In addition, sham tapes will be applied to major postural muscles including the bilateral gluteus medius (i.e., crosses hip joint), quadriceps (i.e., crosses the knee joint), and gastrocnemius (i.e., crosses ankle joint) of the participants.
  Arms: Sham TENS and sham taping

SUMMARY:
Aim: To examine the acute effects of transcutaneous electrical nerve stimulation (TENS) and Kinesio Taping (KT) on lower limb joint proprioception, static standing balance, limits of stability and functional balance performance in community-dwelling older adults.

Design: A one-group experimental study with a repeated-measures design. Sample: 24+ community-dwelling older adults Interventions: TENS and KT, TENS and sham taping, KT and sham TENS, and sham TENS and sham taping (30 minutes each) Major outcomes: Outcomes will be evaluated during each of the intervention conditions. Lower limb joint active repositioning error will be evaluated using a joint position sense test; a force platform will be used to assess the single-leg standing body sway path length and velocity; a functional reach test will give a score that reflects the limits of stability of the participants; and the timed up-and-go test will be used to quantify functional balance performance of the participants.

Anticipated results and significance: It is predicted that both TENS and KT, when applied together, may best improve lower limb joint proprioception and facilitate all balance performances among the community-dwelling older adults. These interventions could be applied in clinical settings to improve joint proprioception and postural control of the elderly people.

ELIGIBILITY:
Inclusion criteria:

* Between 60 and 75 years old
* Able to ambulate independently and safely without using any walking aid
* Able to follow instructions

Exclusion criteria:

* Known unstable medical condition (e.g., uncontrolled hypertension)
* Known sensorimotor or neurological disorders (e.g., stroke and epilepsy)
* Significant musculoskeletal disorder of the lower limbs (e.g., osteoarthritis of the knee)
* Cognitive disorder
* Presence of an implanted electrical device (e.g., cardiac pacemaker)
* Cancer
* A change in skin sensation
* Wound around the lower limb joints
* A recent injury that may affect test performance
* Allergy to adhesive tapes

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Joint active repositioning test error (using goniometry, in degree) | Day 1 to Day 4
  Lower limb joint proprioception test - Joint active repositioning error of the hip, knee and ankle joints of both lower limbs

SECONDARY OUTCOMES:
Center of pressure (COP) sway path length in static single-leg standing (using a force platform, in cm) | Day 1 to Day 4
  Static single-leg standing balance performance - COP sway path length in static single-leg standing
Center of pressure (COP) sway velocity in static single-leg standing (using a force platform, in m/s) | Day 1 to Day 4
  Static single-leg standing balance performance - COP sway velocity in static single-leg standing
Functional Reach Test score (using a cloth measuring tape, in cm) | Day 1 to Day 4
  Limits of stability balance performance - Functional Reach Test score
Timed Up-and-Go Test completion time (using a stop watch, in s) | Day 1 to Day 4
  Functional balance performance - Timed Up-and-Go Test completion time

CONTACTS AND LOCATIONS:
Overall Officials: Shirley SM Fong, PhD, Principal Investigator — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No